CLINICAL TRIAL: NCT01453426
Title: An Open-Label, Parallel-Group, Phase 1 Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of BG00012 in Chinese, Japanese, and Caucasian Adult Healthy Volunteers
Brief Title: Phase 1 Study to Evaluate the PK, Safety, and Tolerability of BG00012 in Chinese, Japanese, and Caucasian Healthy Volunteers
Acronym: 109HV108
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 109HV108
Record Dates: First submitted 2011-10-13; First posted 2011-10-17 (Estimated); Last update posted 2013-09-16 (Estimated); Status verified 2012-05

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Chinese Subjects - Dose 1 BG00012 (Experimental)
  Interventions: Drug: BG00012 Dose 1
- Chinese Subjects - Dose 2 BG00012 (Experimental)
  Interventions: Drug: BG00012 Dose 2
- Japanese Subjects - Dose 1 BG00012 (Experimental)
  Interventions: Drug: BG00012 Dose 1
- Japanese Subjects - Dose 2 BG00012 (Experimental)
  Interventions: Drug: BG00012 Dose 2
- Caucasian Subjects - Dose 1 BG00012 (Experimental)
  Interventions: Drug: BG00012 Dose 1
- Caucasian Subjects - Dose 2 BG00012 (Experimental)
  Interventions: Drug: BG00012 Dose 2

INTERVENTIONS:
Drug: BG00012 Dose 1
  Arms: Caucasian Subjects - Dose 1 BG00012; Chinese Subjects - Dose 1 BG00012; Japanese Subjects - Dose 1 BG00012
Drug: BG00012 Dose 2
  Arms: Caucasian Subjects - Dose 2 BG00012; Chinese Subjects - Dose 2 BG00012; Japanese Subjects - Dose 2 BG00012

SUMMARY:
This is an open-label, parallel-group study to evaluate the PK, safety, and tolerability of two different dose regimens of BG00012 over a 24-hour period to adult Chinese, Japanese, and Caucasian healthy volunteers.

DETAILED DESCRIPTION:
The purpose of this healthy volunteer study is to provide pharmacokinetic and safety data for two different dose regimens of BG00012. The study will evaluate BG00012 administered over a 24-hour period.

The study will be conducted in male and female Chinese, Japanese, and Caucasian healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Must give written informed consent and any authorizations required by local law
* All subjects must practice effective contraception during the study and be willing and able to continue contraception for 30 days after their last dose of study treatment.

Exclusion Criteria:

* History of any clinically significant cardiac, endocrine, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, and renal, or other major disease, as determined by the Investigator.
* History of malignancy (subjects with basal cell carcinoma that has been completely excised prior to study entry remain eligible)
* History of severe allergic or anaphylactic reactions
* Known history of or positive test result for Human Immunodeficiency Virus (HIV)
* Serious infection (e.g., pneumonia, septicemia) within 2 months prior to Screening.
* Female subjects who are pregnant or currently breastfeeding

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2012-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
AUC of BG00012 | First dose to 24 hours
Cmax of BG00012 | First dose to 24 hours

SECONDARY OUTCOMES:
Number of Adverse Events, as a measure of safety and tolerability | Subjects will be followed for the duration of the study, an expected 20 days
Number of Serious Adverse Events, as a measure of safety and tolerability | Subjects will be followed for the duration of the study, an expected 20 days

CONTACTS AND LOCATIONS:
Locations (2):
- Research Site, Melbourne, Victoria, Australia
- Research Site, Hong Kong, Hong Kong, China